CLINICAL TRIAL: NCT05234372
Title: MyVaccineLA/MiVacunaLA: A Mobile Phone Delivered Intervention to Improve COVID-19 Vaccination Behaviors Among Vulnerable Latino Families in Los Angeles
Brief Title: MiVacunaLA: an Intervention to Improve COVID-19 Vaccination Behaviors Among Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Pepperdine University (Other)
Responsible Party: Principal Investigator, Yelba Castellon-Lopez, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 21-000857
Record Dates: First submitted 2022-02-08; First posted 2022-02-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Pandemic
Keywords: vaccination, vulnerable populations, health disparities
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In collaboration with community partners, we designed mivacunaLA as an RCT with a wait-list control group to ensure that all participants could benefit from the educational intervention. The treatment group received the 1 month intervention upon enrollment and the wait-list control received the intervention at month 2 from enrollment. We propose to analyze baseline data for the primary outcomes related to adult caregiver behaviors regarding COVID-19 vaccination for children living in the household for 1 month outcomes, before the control group was exposed to the intervention.
Who Masked: Outcomes Assessor
Masking Description: Participants were informed at enrollment what arm they belonged to. Investigators could see what arm participants were assigned to. Outcome assessors/data analysts was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment received intervention at enrollment (Experimental): Participants received mobile phone delivered intervention at enrollment. The intervention had a duration of 4 weeks. Each week participants received two text messages inviting them to view a short video (Monday) and brief written content (Wed). Each week, the material consisted of a culturally tailored theme related to COVID-19 vaccination. Participants also received information on how to get vaccinated.
  Interventions: Behavioral: mivacunaLA
- Control (Other): Wait-list control. No intervention during month 1. Received the intervention at Month 2. Each week, during the first month, participants received a text with a count down of how many days were left to begin the intervention.
  Interventions: Behavioral: mivacunaLA

INTERVENTIONS:
Behavioral: mivacunaLA — Based on their stated language preference in the baseline survey, eligible participants in the program received a text message or email twice a week (Monday and Wednesday at noon). The short text messages (<160 characters in length) provided a link to a 2-3 min video (Monday) and a short educational content around 500 words (Wednesday). Content was organized by week with the following topics: 1) what is COVID-19 and how COVID-19 vaccines works, 2) COVID-19 vaccine myths and facts, 3) COVID-19 vaccine safety and efficacy in children, and 4) how to obtain COVID-19 vaccines in your community. Every week we provided information about how to get vaccines with links to local vaccine sites & resources.

SUMMARY:
The aim of this study is to determine whether a community-informed, linguistically and culturally tailored educational program delivered via mobile phone is effective in improving vaccination behaviors among Latino families. Thus we evaluate a community-based mobile phone intervention (mivacunaLA) to assess if there is an increase in vaccination rates among 12-17 year old children and willingness to vaccinate 2-11year old children who have not been previously vaccinated who reside in high-risk and low resourced neighborhoods in Los Angeles.

DETAILED DESCRIPTION:
We conducted a community-based randomized clinical trial with a wait list control group among adult Latino parents or caregivers in East and South Los Angeles. Participants completed an online demographic and baseline survey and were randomly assigned to treatment or wait-list control. Based on their preference, participants received a weekly text message or email link twice a week for four weeks (Mon and Wed at noon). Twice a week messages consisted of a short text (<160 characters) linking participants to a 2-3 minute video (Monday) and educational text (around 500 words in length. The material was divided into weekly topics regarding the coronavirus vaccine and other topics relevant to the Latino community. Participants were also directed to reliable websites where they could access additional information and links with instructions on where to get vaccinated. Upon completing the intervention, participants completed a 1-month follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

1. self-identified as Latino/a,
2. were 18 years or older,
3. had at least one unvaccinated child of any age (17 or younger), and
4. had the means to receive messages and review educational material online, such as a text-capable mobile phone with internet access

Exclusion Criteria:

1. Unable to receive information via mobile text or computer.
2. Does not speak English or Spanish.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure: vaccination status among minors 12-17 years | 1 month
  Changes in COVID-19 vaccination status among minors 12-17 years. Have the minor #X 12-17 years old in your household been vaccinated for the coronavirus? 1.Yes, 2.No, 3.Unsure Instrument similar used in the Understanding America Study
Intent to vaccinate children 2-11 yrs old | 1 month
  Change in willingness to vaccinate children 2-11 yrs old. f a vaccine against the coronavirus becomes available for children ages 2-11, do you plan to get them vaccinated?1.Yes, as soon as possible, 2.Yes, but I want to wait and see, 3.No, but I want to wait and see, 4.No, I will not get a coronavirus vaccine for my child, 5.Not sure. Positive answers:1.Yes, as soon as possible, 2.Yes, but I want to wait and see Not positive: 3.No, but I want to wait and see, 4.No, I will not get a coronavirus vaccine for my child, 5.Not sure Instrument adjusted from Understanding America Study.

CONTACTS AND LOCATIONS:
Overall Officials: Yelba M Castellon-Lopez, MD, MS, Principal Investigator — University of California, Los Angeles; Luisa Blanco Raynal, Principal Investigator — Pepperdine University
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Pepperdine University, Malibu, California

IPD SHARING:
Plan to Share IPD: Yes
We have de-identified data available in excel and stata for analysis. Given that our data was collected among a vulnerable population and we did not obtain consent to share PHI at the study onset, with a large immigrant population recruited, our intent is to share de-identified data only through special request by investigators (will need approval by both co-PIs). Sharing of data would be pending approval of our institutional IRB.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will share by special request and pending IRB approval over the next two years.
Access Criteria: Researcher(s) will need to submit an application and it will be reviewed by the co-PIs.